CLINICAL TRIAL: NCT05955911
Title: The Effect of an Acute Exercise Intervention on Alcohol Craving and Alcohol Seeking Behaviors Among Heavy Social Drinkers
Brief Title: Alcohol & Exercise Study
Acronym: Alc-Excr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Jesus Chavarria, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000055296
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Alcohol-Related Disorders
Keywords: Alcohol; Exercise; Heavy Drinkers; Alcohol Craving
MeSH Terms: conditions — Alcohol-Related Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Moderate intensity treadmill walking (40%-59% of heartrate reserve).
  Interventions: Behavioral: Exercise
- Coloring (Other): Coloring in an adult coloring book as a distraction activity
  Interventions: Behavioral: Coloring

INTERVENTIONS:
Behavioral: Exercise — 20 minutes of Moderate intensity (40%-59% heartrate reserve) walking on a treadmill.
  Arms: Exercise
Behavioral: Coloring — 20 minutes of coloring in adult coloring book
  Arms: Coloring

SUMMARY:
The goal of this clinical trial is to learn if exercise can reduce alcohol craving in heavy social alcohol drinkers. The main questions this project aims to answer are 1) compared to a distraction activity (i.e., coloring), will mild-to-moderate intensity exercise (i.e., walking on a treadmill) reduce alcohol craving; 2) compared to a distraction, will mild-to-moderate intensity exercise reduce the amount of consumption of an alcohol-placebo beverage.

DETAILED DESCRIPTION:
Upon arriving to the study, participants will complete baseline measures assessing for the inclusion and exclusion criteria, as well as baseline alcohol craving and subjective response measures. Participants will then be randomly assigned into the active treatment (exercise) or distraction (coloring) condition. After randomization, participants will consume a low-dose alcohol beverage (BAC=0.03g/dL; equivalent to approximately 1 standard alcohol beverage) within five minutes to induce active alcohol craving. 15 minutes post-beverage consumption, participants will complete the alcohol craving and subjective response measures. At 20 minutes post-beverage consumption, participants will begin their randomly assigned 20-minute activity (exercise or coloring). At approximately 12 minutes into the activity (32 minutes post beverage consumption) and immediately after the activity (44 minutes post beverage consumption), the participants will complete the alcohol craving and subjective response measures. Participants will then be given a tray of three 8oz. cups of water and 3 8oz. cups of an alcohol-placebo beverage and will be allowed to drink as much or as little of the beverages as they would like.

ELIGIBILITY:
Inclusion Criteria:

* Heavy social alcohol drinkers (i.e., alcohol drinkers who consume 10-40 standard alcohol beverages per week and participate in 1-5 binge drinking episodes [consume 4+/5+ drinks in a sitting for women/men, respectively]) per week.

Exclusion Criteria:

* Meets DSM-5 diagnostic criteria for a current moderate or severe alcohol use disorder
* Meets DSM-5 diagnostic criteria for a current Moderate or Severe cannabis use disorder
* Endorses daily smoking of tobacco
* Endorses having a current DSM-5 psychiatric disorder
* Endorses having any medical conditions that may interfere with the exercise condition (e.g., knee-replacement, sprained ankle, etc.)
* Has a current level of physical activity that exceeds 20 minutes of moderate-to-vigorous physical activity per day
* Endorses illicit substance use (i.e., use of illicit substances x>2 times in the past year)
* Has self-reported allergies to pineapple juice, cranberry juice, orange juice, &/or tonic water
* Individuals not proficient in reading, writing, or speaking in English
* Women who are trying to conceive or who are pregnant
* Women who are currently breastfeeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Changes in alcohol craving after alcohol prime dose | mid-intervention (32 minutes after prime dose consumption) & post-intervention (44 minutes after prime dose consumption)
  It is expected that the exercise condition will lead to larger reductions in alcohol craving (Alcohol Urge Questionnaire) at the mid- and post-intervention time points as compared to the coloring condition.
Post-intervention alcohol beverage consumption | Post-intervention (approximately 50 minutes after prime dose consumption)
  It is expected that individuals in the exercise condition will consume more of the alcohol-placebo beverage (milliliters of beverage consumed) than individuals in the coloring condition.

SECONDARY OUTCOMES:
Changes in alcohol wanting after alcohol prime dose | mid-intervention (32 minutes after prime dose consumption) & post-intervention (44 minutes after prime dose consumption)
  It is expected that the exercise condition will lead to larger reductions in alcohol wanting (Drug Effects Questionnaire: Want More item) at the mid- and post-intervention time points as compared to the coloring condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Chavarria, Ph.D., Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada